#### CONFIDENTIAL



### CONSENT FORM

# **Participant Identification Number:** Determining the effect of food ordering in Gestational Diabetes Mellitus: a

## Title of Project: Randomized Crossover Study Chief Investigator: Professor Jayne Woodside Study Number: Please initial box 1. I confirm that I have read, or had read to me, and understand the information sheet dated version for the above study. I have had the opportunity to ask questions and these have been answered fully. 2. I understand that my participation is voluntary and I am free to withdraw at any time, without giving any reason and without my legal rights or medical care being affected. 3. I understand the study is being conducted by researchers from Queen's University Belfast and that my personal information will be held securely on University premises and handled in accordance with the Data Protection Act 2018 and General Data Protection Regulations. 4. I understand that data collected as part of this study and may be looked at by authorized individuals from Queen's University Belfast and regulatory authorities where it is relevant to my taking part in this research. I give permission for these individuals to have access to this information. 5. I agree to take part in the above study inclusive of all the procedures mentioned in the participant information sheet. 6. I agree to the Antenatal Clinic I am attending to be informed of my participation in the study. I agree to receive an overall summary of the study results via letter or email once 7. the data has been analysed at the end of the study. 8. I understand that the information I provide may be published as a report. Confidentiality and anonymity will be maintained and it will not be possible to identify me from any publications. 9. I understand that if I withdraw (or lose capacity to consent) during the trial, I agree that data and samples already taken can be retained and used for analysis, but no

Page **1** of **2** IRAS Number: 346910 Version 2.0 11/02/2025

further samples will be collected.

## **CONFIDENTIAL**

| 10. | I agree that study data I provide can be deposited in Queen's University Belfast institutional repository (e.g. PhD thesis) and data produced from this study may be made publicly available, so it can be used for future research and learning. | | from this study may be | |
|---|---|---|---|---|
| 11. | The potential benefits of keeping my blood or other tissues for future research have been explained to me and (please choose <b>one</b> ), | | | |
| | I <u>consent</u> to the storage and use of my blood or other tissues for future research, including genetic analysis, transfer abroad and commercial research. OR | | | |
| | | | | I <u>do not wish</u> my blood or other tissues to be used for any purpose other than this study' |
| | 12. | <b>Optional:</b> I agree to being contacted at a later date by the University and invited to take part in future studies of a similar nature. I understand that I am only agreeing to receive information and I am under no obligation to take part in any future studies. | | |
| If you decide not to consent to being contacted in the future it will not have any influence on your involvement in this particular research study and will not affect any standard of care that you receive. | | | | |
| Name of | Participant (please print) | Signature | <br>Date | |
| Name of Person Taking Consent (please print) | | Signature | Date | |
| Chief Inv | vestigator Contact details: | | | |
| Profess | Professor Jayne Woodside | | | |
| Centre for Public Health | | | | |
| School | of Medicine, Dentistry and B | iomedical Sciences | | |
| Queen's | s University Belfast | | | |
| Institute | e of Clinical Science A | | | |
| Grosve | nor Road | | | |
| Belfast | BT12 6BA | | | |
| Telepho | one: 02890 978942 | | | |
| Email: j.woodside@qub.ac.uk | | | | |

One copy to be kept by the researcher and one copy to be given to the participant.

Page **2** of **2** IRAS Number: 346910 Version 2.0 11/02/2025